CLINICAL TRIAL: NCT02339727
Title: Clinical Trial of the Relation Between Omega-6/Omega-3 Ratio in Formula of Preterm Infants Less Than 1500 Grams and/or Less Than 32 Weeks Gestational Ages and Brunet Lezine Score at 2 Years of Live. Anuvis Study
Brief Title: Omega-6/Omega-3 Ratio and Neural Development in Preterm Infants.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ayham alshweki (Other)
Responsible Party: Sponsor-Investigator, Ayham alshweki, //www.idisantiago.es/, Health Research Institute of Santiago
Organization: Health Research Institute of Santiago (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Ayham alshweki
Record Dates: First submitted 2014-11-14; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Impaired Psychomotor Development
Keywords: Omega-3; Omega-6

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-6/omega-3=2/1 milk formula (Active Comparator): Preterm infants will receive a formulas supplemented with Docosahexaenoic acid and Arachidonic acid with a relationship omega 6/omega 3 = 2/1.
  Interventions: Dietary Supplement: Preterm infants formula
- Omega-6/omega-3=1/1 milk formula (Active Comparator): preterm infants will receive other formulas with Docosahexaenoic acid and Arachidonic acid, but with a ratio of 1/1.
  Interventions: Dietary Supplement: Preterm infants formula

INTERVENTIONS:
Dietary Supplement: Preterm infants formula — The group 1 of children will receive a preterm infants formula supplemented with DHA and ARA with a relationship omega 6/omega 3 = 2/1 during the first 3 months of life. And group 2 will receive other Preterm infants formula very similar, but with a ratio of DHA and AA=1/1 also during the first 3 months of life.

SUMMARY:
It's known that Docosahexaenoic acid DHA and all Polyunsaturated Fatty Acids PUFA are important in neurodevelopment of term and preterm infants. This study tried to determine the utility of a balanced contribution of DHA and Arachidonic acid AA (omega-6/omega-3) in milk formula, with a ratio similar to that found in breastfeeding, equal to 2, in very premature infants less than 1500 grams and / or less than 32 weeks of gestational age. To evaluate values of fatty acids they have in blood and psychomotor development they achieve.

DETAILED DESCRIPTION:
The study took place in a single-center; it is a prospective randomized study of preterm infants less than 1500 grams and/or less than 32 weeks gestational age, admitted to the Neonatal Intensive Care Unit in the University Clinical Hospital of Santiago de Compostela. They were recruited for a period of 14 months (from July 2010 to august 2011) and followed from birth until 2 years of life.

40 children were included and followed in the study. Patients will be assigned randomly into two groups depending on the type of formula they are receiving. The group A of children will receive a formula supplemented with DHA and ARA with a relationship omega 6/omega 3 = 2. And group B will receive other formula with DHA and ARA, but with a ratio of 1/1.

The classification of group A and B was made by simple random way; one birth in every group, continuously.

Implementation of breastfeeding will be promoted and will be fortified after 7 days of life, when the total amount of breast milk will be more than 1/2 of the total.

When breastfeeding will be insufficient or nonexistent, special formulas for premature babies will be given

During the follow-up of patients, will be measured:

1. - Levels of fatty acids in blood in the first week of life, 3 months, 6 months and 12 months.The determination will be carried out in collaboration with the Hospital de Cruces, Bilbao, Spain.
2. - Evaluation of psychomotor development by Brunet-Lezine scale at 2 years of corrected age.

ELIGIBILITY:
Inclusion Criteria:

Living infants who were less than 1500 grams and/or less than 32 weeks gestational age, and whose parents accepted and subscribed the informed consent

Exclusion Criteria:

* Preterm infants with any malformation or deformation.
* Extreme preterm infants with gestational age less than 25 weeks.
* Infants whose parents couldn't follow up their children in our study center.
* Preterm infants who had a severe intra ventricular hemorrhage (more than grade 2).
* Premature infants who had severe periventricular leukomalacia (more than grade 2) because the latest two conditions can affect neurodevelopment.
* Finally, we excluded neonates who don't need supplementary milk nutrition, i.e. children with breastfeeding only.

Ages: 1 Minute to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Levels of fatty acids in blood | from July 2010 to august 2012 (from the birth to 1 years old)
  Levels of fatty acids in blood in the first week of life, 3 months, 6 months and 12 months of live

SECONDARY OUTCOMES:
Psychomotor development | from september 2012 to november 2013 (at two years of corrected age)
  Evaluation of psychomotor development by making Brunet-Lezine scale at 2 years of corrected age.